CLINICAL TRIAL: NCT03475771
Title: Retrospective Evaluation of Thrombo-embolic Complication in Pelvic Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MTEVbassin
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Venous Thromboembolism; Pelvic Fracture
MeSH Terms: conditions — Venous Thromboembolism; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pelvic fracture are very often treated by surgery ; however there are a high level of thrombotic risk during the surgery (venous thrombo embolic events represent about 10% to 50%.

The aim of our study is to report the number of these events and identify the risk factor associated to these events regarding Greenfield Risk Assessment Profile .

ELIGIBILITY:
Inclusion Criteria:

* indication to pelvic fracture surgery
* age above 18 years

Exclusion Criteria:

* pelvic fracture without surgery indication.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients admitted in GHPSJ orthopedy yard between december 2014 and january 2017
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
number of venous thrombo-embolic events | Month 1

CONTACTS AND LOCATIONS:
Overall Officials: BONHOMME Stéphanie, MD, Principal Investigator — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France